CLINICAL TRIAL: NCT07287163
Title: Open Label Extension Clinical Trial of Vormatrigine in Adult Patients With Epilepsy
Brief Title: Clinical Trial of Vormatrigine in Adult Patients With Epilepsy
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRAX-628-323
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy, Tonic-Clonic; Focal Seizure; Primary Generalized Seizure
Keywords: epilepsy; tonic-clonic; seizure; focal
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label 30 mg/day vormatrogine for up to 2 years (Experimental): Participants who meet all eligibility criteria will receive 30 mg of vormatrogine for up to 2 years.
  Interventions: Drug: vormatrogine

INTERVENTIONS:
Drug: vormatrogine — Once daily oral

SUMMARY:
Open Label Extension Clinical Trial of Vormatrigine in Adult Patients with Epilepsy

DETAILED DESCRIPTION:
An open label extension clinical trial to assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures.

ELIGIBILITY:
Inclusion Criteria:

* Participant who completed an eligible clinical trial (unless agreed by the sponsor medical monitor), including PRAX-628-212, PRAX-628-321 or other vormatrigine trials, or participant who has received vormatrigine outside of an eligible clinical trial (such as an expanded access program)
* Participant who had adequate seizure diary and vormatrigine adherence and had been otherwise adherent to the study procedures in the opinion of the investigator unless deemed unacceptable by sponsor

Exclusion Criteria:

* Participant who withdrew or discontinued treatment from the treatment period of an eligible clinical trial unless deemed acceptable by the sponsor
* Participant who plans to enter another interventional investigational study or is on any prohibited medication
* Participant who is pregnant, lactating or planning to become pregnant
* Participant who is ineligible for the extension clinical trial in the view of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Incidence and severity of TEAEs including discontinuation of study drug due to TEAEs
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Change in tympanic temperature in Celsius
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Change in heart rate in beats per minute
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Change in blood pressure in mm/Hg
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Change in respiratory rate in breaths per minute
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  The principal investigator (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.
To assess the safety and tolerability of vormatrigine in adults with focal or primary generalized tonic-clonic seizures | Up to 2 years
  Incidence of clinically significant ECG abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (20):
- United States (9):
  - Praxis Research Site, Miami Lakes, Florida
  - Praxis Research Site, Naples, Florida
  - Praxis Research Site, Lafayette, Louisiana
  - Praxis Research Site, Bethesda, Maryland
  - Praxis Research Site, Chesterfield, Missouri
  - Praxis Research Site, Amherst, New York
  - Praxis Research Site, Middletown, New York
  - Praxis Research Site, El Paso, Texas
  - Praxis Research Site, Houston, Texas
- Germany (2):
  - Praxis Research Site, Bielefeld
  - Praxis Research Site, Tübingen
- Italy (2):
  - Praxis Research Site, Milan
  - Praxis Research Site, Pavia
- Poland (2):
  - Praxis Research Site, Bydgoszcz
  - Praxis Research Site, Katowice
- Spain (5):
  - Praxis Research Site, Barcelona
  - Praxis Research Site, Madrid
  - Praxis Research Site, Málaga
  - Praxis Research Site, Terrassa
  - Praxis Research Site, Valencia